CLINICAL TRIAL: NCT03782025
Title: Effect of Vitamin K in Critically Ill Patients With Spontaneously Increased Pro-thrombin Time Measured With Routine Coagulation Tests and Advanced Coagulation- and Vitamin K-assays
Brief Title: Effect of Vitamin K in Critically Ill Patients
Acronym: VITAKOAG
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Thomas Kander, Consultant, Region Skane
Other Study IDs: VITAKOAG
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Coagulation Factor Deficiency; Coagulopathy, Consumption; Vitamin K Deficiency
MeSH Terms: conditions — Disseminated Intravascular Coagulation; Vitamin K Deficiency | interventions — Vitamin K 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be centrifuged and stored in -80 degrees C in anticipation of batch analysis of coagulation factor- and vitamin K-analyses. There will be no DNA analysis. All blood samples will be destroyed after the mentioned analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with increased PK-INR: Critically ill patients with spontaneously increased prothrombin complex (PK-INR) who are given phytomenadione intravenously at the discretion of the treating physician
  Interventions: Drug: Phytomenadione

INTERVENTIONS:
Drug: Phytomenadione — Blood samples will be taken before and after intravenously prescribed phytomenadione is given. Phytomenadione will be given independently of this study.

SUMMARY:
Critically ill patients with spontaneously prolonged pro-thrombin time, where administration of intravenous administration of phytomenadione (vitamin K) has been ordered by the treating physician will be identified. After signed informed consent baseline samples will be collected. Phytomenadione will be given and 24 hours after administration new blood samples will be collected. Several different advanced coagulation and vitamin K-assays will be performed before and 24 hours after vitamin K administration.

DETAILED DESCRIPTION:
Vitamin K-deficiency is common in the peri-operative and intensive care setting. It is often seen in patients with prolonged prothrombin complex (PK-INR). A prolonged (PK-INR) is sometimes treated with intravenous vitamin K, even in non-warfarin treated or non-liver failure patients. Despite the development of this practice the knowledge about how intravenously given vitamin K affects routine coagulation status and other advanced laboratory coagulations assays is rare.

The aim of this study is to investigate the effects of intravenously administered vitamin K on routine coagulation status and on advanced coagulation and vitamin K-assays in post-operative- and critically ill patients with prolonged PK-INR.

Patients with spontaneously prolonged PK-INR are routinely given intravenous vitamin K but it is largely unknown how this procedure affects the included coagulation assays. This research project may contribute to increased knowledge concerning effects of intravenously given vitamin K in critical ill patients with spontaneous coagulopathies. Since spontaneous coagulopathy is frequently occurring in critically ill and postoperative patients due to various underlying conditions and current evidence for vitamin K administration is based on scarce evidence more research in this area is motivated.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients at the postoperative care unit or at the intensive care unit with a prothrombin complex (PK-INR) > 1.2 during office hours who are ordered parenteral phytomenadione 10 mg will be eligible for inclusion

Exclusion Criteria:

* Warfarin treatment
* Treatment with novel oral anticoagulants
* Hepatocellular carcinoma
* Liver resection within 6 months
* Known pre-existing coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients at the postoperative care unit or at the intensive care unit with a prothrombin complex (PK-INR) > 1.2 during office hours who are ordered parenteral phytomenadione 10 mg will be eligible for inclusion
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change in prothrombin complex (PK-INR) | Before and 24 hours after given phytomenadione
  Prothrombin complex (PK-INR) with Owren and Quick reagents

SECONDARY OUTCOMES:
Change in concentration of coagulation factors II, VII, IX and X in plasma | Before and 24 hours after given phytomenadione
Change in concentration of PIVKA-II in plasma | Before and 24 hours after given phytomenadione
  Protein Induced by Vitamin K Absence or antagonism for factor II (PIVKA-II)
Change in concentration of protein C and S in plasma | Before and 24 hours after given phytomenadione
Change in concentration of dp-ucMGP in plasma | Before and 24 hours after given phytomenadione
  Dephospho-uncarboxylated Matrix Gla Protein (dp-ucMGP)
Change in thrombin generation assay in plasma | Before and 24 hours after given phytomenadione
Change in thromboelastometry assay in whole blood | Before and 24 hours after given phytomenadione
  Thromboelastometry using ROTEM with tissue factor activation (EXTEM reagent)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kander, Ass. Prof., Principal Investigator — Skane University Hospital
Locations (2):
- Sweden (2):
  - Intensive and perioperative care. Skåne University Hospital. Lund, Lund, Skåne County
  - Skåne University Hospital, Lund, Skåne County

IPD SHARING:
Plan to Share IPD: No